CLINICAL TRIAL: NCT06899152
Title: HepQuant: Pilot Study to Assess the Role of Blood-based Biomarkers and Quantitative MR Imaging for Patients Receiving Radiation Therapy for Liver Cancer
Brief Title: HepQuant: Study to Assess the Role of Blood-based Biomarkers and Quantitative MR Imaging for Patients Receiving Radiation Therapy for Liver Cancer
Acronym: HepQuant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: HepQuant, LLC (Industry); Perspectum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-16581
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Hepatocellular Cancer; Cholangiocarcinoma; Liver Metastases
Keywords: Blood-based biomarkers; Quantitative MR imaging; Radiotherapy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Multiparametric MRI scans and HepQuant Duo Test (Experimental)
  Interventions: Diagnostic Test: HepQuant DuO; Other: Multiparametric MRI Scans
- Multiparametric MRI scans only (Active Comparator)
  Interventions: Other: Multiparametric MRI Scans

INTERVENTIONS:
Diagnostic Test: HepQuant DuO — HepQuant DuO is a quantitative liver function test. It assesses cholate uptake, a liver specific function. Cholate is a naturally occurring substance that is cleared by the liver. Cholate uptake reflects the health of liver cells.
  Arms: Multiparametric MRI scans and HepQuant Duo Test
Other: Multiparametric MRI Scans — Standard of care

SUMMARY:
This is a pilot and feasibility study assessing the role of quantitative multiparametric MRI and blood-based biomarkers for the measurement of liver function in patients receiving radiation therapy for liver cancer, including hepatocellular carcinoma (HCC), cholangiocarcinoma, or liver metastases regardless of primary histology, that are undergoing photon radiation either in the de-novo or re-irradiation setting. The goal of this study is to prospectively evaluate the feasibility of using quantitative multiparametric MRI to monitor liver function at baseline and following liver radiation therapy.

DETAILED DESCRIPTION:
Historically, the role of fractionated liver radiation therapy (RT) has been limited because of the potential for developing fatal radiation-induced liver disease (RILD), particularly in patients who already have poor liver function due to cirrhosis. Classic RILD generally occurs within 4 months following radiotherapy to the liver and consists of symptoms including fatigue, right upper quadrant pain, ascites, anicteric hepatomegaly, and elevation of liver enzymes especially alkaline phosphatase.

Technical advances in the delivery of RT, particularly using stereotactic body radiotherapy (SBRT) and proton therapy with respiratory gating and image guidance, have facilitated the safe use of radiation dose escalation in unresectable liver cancers. SBRT is a promising and attractive option for HCC patients with cirrhosis. Previous reported experiences have been largely kept to Child-Pugh (CP) A patients with significant liver reserves. The 1 to 2-year local control rate for CP A patients with early-stage tumor have generally been reported around 80-90%. Toxicities rates have also been acceptable with no classic RILD or grade 4 or 5 treatment related toxicities seen 3 months after SBRT. This impressive toxicity result is likely due to keeping with strict dosimetric constraints for the normal liver tissue. Dosimetric parameters reported in literature indicated mean liver disease (MLD) and V20 to be a significant predictor of RILD and elevated liver enzymes in CP A patients with primary HCC.

While there are no overt liver toxicities in CP A patients with primary liver cancer, 10 to 30% of patients will experience a decline in liver function 3 months after SBRT even without disease progression based on the referenced literature. Pre-treatment CP A6 has an increased risk of liver function decline when compared to CP A5. In addition, the tumor volume was also a significant predictor of liver function decline after SBRT.

Patients with CP B or C and primary HCC are more likely to experience liver toxicities as defined by worsening liver function. Dosimetric parameters to predict for fatal RILD for this group has also remained elusive. Yet, it is this particular group of patients that have the worst outcome due to limited treatment options as a result of poor liver reserve to tolerate currently available treatments. The median survival for patients with Child-Pugh B or C HCC treated with best supportive care or sorafenib is approximately 4-5 months according to the literature. Limited institutional experiences have shown that local treatment of these patients with SBRT can potentially improve survival; however, this also comes at a cost of significant potential toxicity. Current reported data are limited, but they do show that patients can experience liver function decline as early as 3 months.

The published experience with SBRT in the treatment of HCC clearly demonstrates a relationship of the underlying degree of hepatic impairment to risk for liver toxicity. However, the data also clearly demonstrate that CP class or score is insufficient to define risk or to monitor treatment effects. The proposed study will use blood-based biomarkers coupled with quantitative imaging (LiverMultiScan™) to fully characterize the effect of SBRT on the liver and the liver cancer.

In vivo Multiparametric MR imaging (mpMRI) is well established at quantifying measures of liver health in patients with liver disease and pre-clinical models of liver disease. In patients with pre-existing/co-existing parenchymal liver disease and liver tumors (primary or secondary), mpMRI can be used to assess the health of the parenchyma and the anatomical and tissue characteristics of the tumor. This allows for decision-making to be based on the health of the liver and the resectability of the tumor. Initial data suggests that this approach can predict which operations will carry higher risk and cost, measured by length of stay in hospital after surgery.

A more sensitive laboratory measure that is currently available in the U.S. as a Laboratory Developed Test (LDT) to measure liver function and will be used in this study as an investigational assay, is the HepQuant DuO test. It measures cholate hepatic uptake from portal circulation and estimates hepatic uptake from systemic circulation to calculate degree of portosystemic shunting as well as hepatic function using the disease severity index (DSI). Both of these measures have been shown to correlate with severity of chronic liver disease and in studies detected and measured the severity and progression of disease and the response to treatments. The HepQuant DuO test is done by oral administration of unconjugated cholate and collection of two serum samples up to 60 minutes after administration. HepQuant DuO may offer a unique capability to assesses liver functional impairment across the spectrum of injury and fibrosis in patients undergoing radiation therapy to better predict clinical outcomes and risk of liver function deterioration.

ELIGIBILITY:
The following criteria must be met for subjects to be considered for the trial. Additional exclusion criteria must be met for subjects interested in the HepQuant subset of the trial. The first 20 qualifying subjects will be enrolled for the additional HepQuant test.

Inclusion Criteria:

* Age > 18
* Patient has the psychological ability and general health needed to provide informed consent, completion of study requirements, and required follow-up
* Patient provides study-specific informed consent prior to study entry
* All primary histologies (Hepatocellular carcinoma or Cholangiocarcinoma) as well as hepatic metastases are eligible
* Prior history of radiation therapy (external beam or radioembolization) is allowed, with no limit to the number of prior courses of radiation therapy
* Any number of lesions (with no size limit) of pathologically documented (histologically or cytologically) or radiographically proven tumor/metastasis that are being targeted
* Prior history of liver resection, transarterial chemoembolization (TACE), or ablation are allowed with no restriction on number of prior therapies, or time from current study registration
* Prior history of chemotherapy, immunotherapy, or targeted biological therapy is allowed
* Concurrent enrollment on other prospective registry or treatment intention trials is allowed

Exclusion Criteria:

* Pregnant or breast-feeding females
* Subjects with history of claustrophobia impacting ability to perform MRI during the study
* Subjects who fulfill any of the contraindications for MRI; examples include any ferromagnetic material, any metallic shrapnel or fragments or implanted electronic devices contained within the body or metal-containing tattoos
* Unable to participate in MR assessments due to physical limitations of equipment tolerances (MRI bore size and/or weight limit)
* Any person unable to lie still within the environment of the MRI scanner or maintain a breath hold for the required period to acquire images

Exclusion criteria for HepQuant SHUNT DuO testing ONLY:

* Known history or suspected hypersensitivity to human serum albumin, or its preparations
* Subjects with extensive resection of large segments of small intestine (short gut) or severe gastroparesis (e.g., diabetic or medication-induced gastroparesis)
* Subjects on either a non-selective beta blocker (propranolol, nadolol), or an angiotensin converting enzyme (ACE) inhibitor, or angiotensin receptor blocker (ARB) who are unwilling or unable to delay taking their normal dose the morning of their testing
* Subjects who are allergic to any ingredient in the formulations or components in the HepQuant SHUNT DuO kit including the human serum albumin (HSA) or cholate compounds (theoretical - none yet reported)
* Subjects unwilling or unable to fast for at least 5 hours. Fasting means no intake of food or food supplements, including fiber preparations or biosimilars; or any preparations or resins (cholestyramine, colestipol, colesevelam) that might act within the gut lumen to bind the orally administered d4-cholate in the HepQuant test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Quantitative MRI | Approximately 3 months
  Feasibility will be determined by assessing the proportion/percentage of participants who complete at least 2 quantitative multiparametric MRI scans following study enrollment. The proportion/percentage of patients will be summarized by study arm using basic descriptive statistics and a Clopper-Pearson 95% exact confidence interval will be determined.

SECONDARY OUTCOMES:
Change in Disease Severity Index (DSI) score | From baseline to 3 months post-SBRT
  Change in DSI scores from baseline will be evaluated using the HepQuant DuO test. The HepQuant DuO test measures the liver's ability to clear cholate from the blood using the Disease Severity Index (DSI). The DSI is a single score calculation that incorporates measures of both hepatocyte function and portal circulation and is calculated by indexing a patient's hepatic filtration rate (HFR) against maximum HFR and generates a liver DSI score ranging from 0 (no hepatic disease) to 50 (severe hepatic disease) such that increased DSI scores are correlated with worsening liver function and disease severity and progression. For purposes of this study change in DSI score from baseline will be summarized using basic descriptive statistics and will be examined using a Wilcoxon Sign rank test.
Predictive ability of LiverMultiScan | 6 months post-SBRT
  The ability of the LiverMultiScan to predict the risk of non-classic RILD will be evaluated. The pre-SBRT liver health assessment score will be calculated by measuring the Future Liver Remnant volume outside the 50% radiation isodose line weighted by the liver cT1 value. MRI images will be post-processed using LiverMultiScan, which provides a multiparametric quantitative map of a region of interest in the liver including characterization of the underlying liver fibroinflammation as reported by a corrected T1 (cT1) value, which will be measured and reported in milliseconds (ms). The likelihood of non-classic RILD based on the cT1 value will be assessed using multivariable logistic regression.
  Non-classic RILD will be defined as either worsening of Child-Pugh Score by >=2 points (overall range: 5-15 points) at 6 months following SBRT or an elevated aminotransferase (ALT or AST) level > 5 times the upper limit of normal or baseline value within 90 days of completion of SBRT.
Change in Total Liver Volume | From baseline to 3 months, 6 months, 9 months and 12 months post-SBRT
  Change in total liver volume from pre-SBRT treatment at baseline will be evaluated using Gd-EOB-DTPA enhanced MRI of the abdomen at the specified timeframes to assess the impact of radiotherapy. Mean changes in total liver volume (in mL or cm^3) will be assessed using the MRI software image analysis and summarized by study arm and data will be analyzed using linear mixed-effects models. Increases in liver volume are correlated to more favorable outcomes.
Change in volume of non-irradiated and irradiated liver lobes | From baseline to 3 months, 6 months, 9 months and 12 months post-SBRT
  Change in volume of non-irradiated and irradiated liver lobes, from pre-SBRT treatment at baseline will be evaluated using Gd-EOB-DTPA enhanced MRI of the abdomen at the specified timeframes to assess the impact of radiotherapy. Mean changes in the volume of non-irradiated and irradiate lobes (in mL or cm^3) will be assessed using the MRI software image analysis and summarized by study arm and data will be analyzed using linear mixed-effects models. Increases in liver lobe volume are correlated to more favorable outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Kabarriti, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell AH, Clyde C, Wasserman TH, Turner SS, Rotman M. Accelerated hyperfractionated hepatic irradiation in the management of patients with liver metastases: results of the RTOG dose escalating protocol. Int J Radiat Oncol Biol Phys. 1993 Sep 1;27(1):117-23. doi: 10.1016/0360-3016(93)90428-x. PMID 8365932
- [Background] Ben-Josef E, Lawrence TS. Radiotherapy for unresectable hepatic malignancies. Semin Radiat Oncol. 2005 Oct;15(4):273-8. doi: 10.1016/j.semradonc.2005.04.006. PMID 16183481
- [Background] Dawson LA, Guha C. Hepatocellular carcinoma: radiation therapy. Cancer J. 2008 Mar-Apr;14(2):111-6. doi: 10.1097/PPO.0b013e31816a0e80. PMID 18391616
- [Background] Tse RV, Guha C, Dawson LA. Conformal radiotherapy for hepatocellular carcinoma. Crit Rev Oncol Hematol. 2008 Aug;67(2):113-23. doi: 10.1016/j.critrevonc.2008.01.005. Epub 2008 Mar 4. PMID 18308583
- [Background] Ohri N, Tome WA, Mendez Romero A, Miften M, Ten Haken RK, Dawson LA, Grimm J, Yorke E, Jackson A. Local Control After Stereotactic Body Radiation Therapy for Liver Tumors. Int J Radiat Oncol Biol Phys. 2021 May 1;110(1):188-195. doi: 10.1016/j.ijrobp.2017.12.288. Epub 2018 Jan 6. PMID 29395629
- [Background] Tse RV, Hawkins M, Lockwood G, Kim JJ, Cummings B, Knox J, Sherman M, Dawson LA. Phase I study of individualized stereotactic body radiotherapy for hepatocellular carcinoma and intrahepatic cholangiocarcinoma. J Clin Oncol. 2008 Feb 1;26(4):657-64. doi: 10.1200/JCO.2007.14.3529. Epub 2008 Jan 2. PMID 18172187
- [Background] Miften M, Vinogradskiy Y, Moiseenko V, Grimm J, Yorke E, Jackson A, Tome WA, Ten Haken RK, Ohri N, Mendez Romero A, Goodman KA, Marks LB, Kavanagh B, Dawson LA. Radiation Dose-Volume Effects for Liver SBRT. Int J Radiat Oncol Biol Phys. 2021 May 1;110(1):196-205. doi: 10.1016/j.ijrobp.2017.12.290. Epub 2018 Jan 6. PMID 29482870
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Su TS, Luo R, Liang P, Cheng T, Zhou Y, Huang Y. A prospective cohort study of hepatic toxicity after stereotactic body radiation therapy for hepatocellular carcinoma. Radiother Oncol. 2018 Oct;129(1):136-142. doi: 10.1016/j.radonc.2018.02.031. Epub 2018 Mar 13. PMID 29548558
- [Background] Hasan S, Thai N, Uemura T, Kudithipudi V, Renz P, Abel S, Kirichenko AV. Hepatocellular carcinoma with child Pugh-A Cirrhosis treated with stereotactic body radiotherapy. World J Gastrointest Surg. 2017 Dec 27;9(12):256-263. doi: 10.4240/wjgs.v9.i12.256. PMID 29359031
- [Background] Nabavizadeh N, Waller JG, Fain R 3rd, Chen Y, Degnin CR, Elliott DA, Mullins BT, Patel IA, Dyer BA, Fakhoury K, Naugler WE, Farsad K, Tanyi JA, Fuss M, Thomas CR Jr, Hung AY. Safety and Efficacy of Accelerated Hypofractionation and Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma Patients With Varying Degrees of Hepatic Impairment. Int J Radiat Oncol Biol Phys. 2018 Mar 1;100(3):577-585. doi: 10.1016/j.ijrobp.2017.11.030. Epub 2017 Nov 27. PMID 29413273
- [Background] Cheng JC, Wu JK, Huang CM, Huang DY, Cheng SH, Lin YM, Jian JJ, Yang PS, Chuang VP, Huang AT. Radiation-induced liver disease after radiotherapy for hepatocellular carcinoma: clinical manifestation and dosimetric description. Radiother Oncol. 2002 Apr;63(1):41-5. doi: 10.1016/s0167-8140(02)00061-0. PMID 12065102
- [Background] Hollebecque A, Cattan S, Romano O, Sergent G, Mourad A, Louvet A, Dharancy S, Boleslawski E, Truant S, Pruvot FR, Hebbar M, Ernst O, Mathurin P. Safety and efficacy of sorafenib in hepatocellular carcinoma: the impact of the Child-Pugh score. Aliment Pharmacol Ther. 2011 Nov;34(10):1193-201. doi: 10.1111/j.1365-2036.2011.04860.x. Epub 2011 Sep 29. PMID 21958438
- [Background] Marrero, J., et al. Global Investigation of Therapeutic Decisions in Hepatocellular Carcinoma and of its Treatment with Sorafenib (GIDEON) second interim analysis in more than 1,500 patients: Clinical findings in patients with liver dysfunction. in ASCO Annual Meeting Proceedings. 2011.
- [Background] Cardenes HR, Price TR, Perkins SM, Maluccio M, Kwo P, Breen TE, Henderson MA, Schefter TE, Tudor K, Deluca J, Johnstone PA. Phase I feasibility trial of stereotactic body radiation therapy for primary hepatocellular carcinoma. Clin Transl Oncol. 2010 Mar;12(3):218-25. doi: 10.1007/s12094-010-0492-x. PMID 20231127
- [Background] Culleton S, Jiang H, Haddad CR, Kim J, Brierley J, Brade A, Ringash J, Dawson LA. Outcomes following definitive stereotactic body radiotherapy for patients with Child-Pugh B or C hepatocellular carcinoma. Radiother Oncol. 2014 Jun;111(3):412-7. doi: 10.1016/j.radonc.2014.05.002. Epub 2014 Jun 3. PMID 24906626
- [Background] Weiner AA, Olsen J, Ma D, Dyk P, DeWees T, Myerson RJ, Parikh P. Stereotactic body radiotherapy for primary hepatic malignancies - Report of a phase I/II institutional study. Radiother Oncol. 2016 Oct;121(1):79-85. doi: 10.1016/j.radonc.2016.07.020. Epub 2016 Aug 23. PMID 27566894
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Jayaswal ANA, Levick C, Collier J, Tunnicliffe EM, Kelly MD, Neubauer S, Barnes E, Pavlides M. Liver cT1 decreases following direct-acting antiviral therapy in patients with chronic hepatitis C virus. Abdom Radiol (NY). 2021 May;46(5):1947-1957. doi: 10.1007/s00261-020-02860-5. Epub 2020 Nov 28. PMID 33247768
- [Background] Janowski K, Shumbayawonda E, Dennis A, Kelly M, Bachtiar V, DeBrota D, Langford C, Thomaides-Brears H, Pronicki M, Grajkowska W, Wozniak M, Pawliszak P, Chelstowska S, Jurkiewicz E, Banerjee R, Socha P. Multiparametric MRI as a Noninvasive Monitoring Tool for Children With Autoimmune Hepatitis. J Pediatr Gastroenterol Nutr. 2021 Jan 1;72(1):108-114. doi: 10.1097/MPG.0000000000002930. PMID 32925554
- [Background] Mole DJ, Fallowfield JA, Sherif AE, Kendall T, Semple S, Kelly M, Ridgway G, Connell JJ, McGonigle J, Banerjee R, Brady JM, Zheng X, Hughes M, Neyton L, McClintock J, Tucker G, Nailon H, Patel D, Wackett A, Steven M, Welsh F, Rees M; HepaT1ca Study Group. Quantitative magnetic resonance imaging predicts individual future liver performance after liver resection for cancer. PLoS One. 2020 Dec 2;15(12):e0238568. doi: 10.1371/journal.pone.0238568. eCollection 2020. PMID 33264327
- [Background] Sethi P, Thavanesan N, Welsh FK, Connell J, Pickles E, Kelly M, Fallowfield JA, Kendall TJ, Mole DJ, Rees M. Quantitative multiparametric MRI allows safe surgical planning in patients undergoing liver resection for colorectal liver metastases: report of two patients. BJR Case Rep. 2021 Jan 12;7(3):20200172. doi: 10.1259/bjrcr.20200172. eCollection 2021 May 1. PMID 34131498
- [Background] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Lauriski S, Curto TM, Stoddard A, Wright EC; HALT-C Trial Group. Quantitative liver function tests improve the prediction of clinical outcomes in chronic hepatitis C: results from the Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial. Hepatology. 2012 Apr;55(4):1019-29. doi: 10.1002/hep.24752. Epub 2012 Mar 1. PMID 22030902
- [Background] Burton JR Jr, Helmke S, Lauriski S, Kittelson J, Everson GT. The within-individual reproducibility of the disease severity index from the HepQuant SHUNT test of liver function and physiology. Transl Res. 2021 Jul;233:5-15. doi: 10.1016/j.trsl.2020.12.010. Epub 2021 Jan 2. PMID 33400995